CLINICAL TRIAL: NCT05929443
Title: Feasibility of a Theory-based Benzodiazepines Deprescribing Intervention in Belgian Nursing Homes: the END-IT Study
Brief Title: Benzodiazepines Deprescribing in Nursing Homes: Intervention Feasibility
Acronym: END-IT NH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Collaborators: EBPracticenet (Unknown); Fonds National de la Recherche scientifique (FNRS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLIP/2023/02
Record Dates: First submitted 2023-05-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Benzodiazepines Deprescribing
Keywords: Benzodiazepines; Deprescribing; Long-term care; Older adults
MeSH Terms: interventions — Nursing Homes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- END-IT intervention for nursing homes (Experimental): This complex intervention, implemented at the level of the nursing home, encompasses process and goals setting, education for healthcare providers, environmental adaptations, audit and feedback on benzodiazepine use, use of an educational leaflet for residents and relatives, and multidisciplinary work.
  Interventions: Other: END-IT intervention for nursing homes
- Control (No Intervention): Usual care. Nursing homes allocated to this study arm will access intervention material at the end of the study.

INTERVENTIONS:
Other: END-IT intervention for nursing homes — Complex intervention, as described in the arm/group descriptions
  Arms: END-IT intervention for nursing homes

SUMMARY:
The goal of this feasibility study is to evaluate the feasibility of a complex intervention towards benzodiazepines and Z-drugs deprescribing in older adults living in the Belgian nursing home setting.

The main questions it aims to answer are:

* Is the intervention we developped feasible
* To what extent will the intervention be implemented in nursing homes
* To what extent is the design of the recruitment and data collection process feasible and acceptable for all participants

Participants will benefit from a complex intervention implemented at the level of the nursing home, encompassing process and goals setting, healthcare providers education, environmental adaptations, audit and feedback on benzodiazepines use, use of educational leaflet with residents and relatives, and multidisciplinary work.

Researchers will compare this intervention to usual care, to see if the intervention is feasible, and to gather first data on intervention effectiveness in benzodiazepines deprescriping.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old and older
* Taking at least one benzodiazepine or Z-drug for 4 weeks or more

Exclusion Criteria:

* Unability to communicate in French
* Palliative care
* Ongoing benzodiazepine withdrawal
* Ongoing alcohol withdrawal
* Severe anxiety
* Severe depression

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Nursing homes' adherence to the intervention | Assessed at 6 months
  has the intervention been implemented as intended, e.g. global number of implemented intervention components
Healthcare providers responsiveness to the intervention | Assessed at 6 months
  has far did they respond to the intervention, and how far have them been engaged by the intervention, e.g level of attendance to education session for healthcare providers
nursing home residents' responsiveness to the intervention | Assessed at 6 months
  has far did they respond to the intervention, and how far have them been engaged by the intervention
Feasibility of the recruitment process | At 6 months
  The feasibility of the recruitment will be assessed through the ratio between included residents and residents contacted for participation.
Feasibility of the data collection process | At 6 months
  Data collection process will be assessed through the quality of collected data (rate of missing data)

SECONDARY OUTCOMES:
Contextual factors at the level of of the nursing home | Baseline
  Use of a questionnaire to assess factors that could explain potential differences in intervention implementation between nursing homes
Contextual factors at the level of the nursing home resident | Baseline
  Use of a questionnaire to assess factors that could explain potential differences in intervention implementation between nursing home residents
Intervention mechanisms of impact | At baseline
  Use of a questionnaire to assess intervention mechanisms of impact, in relation with how the intervention is supposed to have its impact
Intervention mechanisms of impact | At 3 months
  Use of a questionnaire to assess intervention mechanisms of impact, in relation with how the intervention is supposed to have its impact.
Intervention mechanisms of impact | At 6 months
  Use of a questionnaire to assess intervention mechanisms of impact, in relation with how the intervention is supposed to have its impact.
Exploratory benzodiazepine deprescribing rate analysis | At 3 months
  Defined as either a complete benzodiazepine/Z-drug cessation, or a dose reduction
Exploratory benzodiazepine deprescribing rate analysis | At 6 months
  Defined as either a complete benzodiazepine/Z-drug cessation, or a dose reduction

CONTACTS AND LOCATIONS:
Overall Officials: Anne Spinewine, PhD, Principal Investigator — UCLouvain / Louvain Drug Research Institute / Clinical pharmacy research group
Locations (1):
- UCLouvain, Woluwe-Saint-Lambert, Belgium

IPD SHARING:
Plan to Share IPD: No
Only publishable project data relating to the main analysis and research output will be shared on a data repository after an embargo period of two years after June 2024. All relevant documentation necessary to facilitate data re-use will be shared along with the datasets.

REFERENCES:
- [Derived] Evrard P, Chevallereau T, Aikpitanyi J, Petein C, Tubeuf S, Henrard S, Spinewine A. Feasibility of a theory-based intervention towards benzodiazepine deprescribing in Belgian nursing homes: protocol of the END-IT NH cluster-randomised controlled trial. BMJ Open. 2024 Oct 22;14(10):e085435. doi: 10.1136/bmjopen-2024-085435. PMID 39438099